CLINICAL TRIAL: NCT00653003
Title: To Compare the Relative Bioavailability of Leflunomide 20mg Tablets (Kali) With That of ARAVA 20mg Tablets(Aventis) Under Fed Conditions
Brief Title: Bioavailability Study of Leflunomide Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Dr. Alfred Elvin/Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2004-704
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: Bioequivalence, Leflunomide, fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Kali formulated product under fed conditions
  Interventions: Drug: Leflunomide
- B (Active Comparator): Subjects received Aventis formulated products under fed conditions
  Interventions: Drug: ARAVA

INTERVENTIONS:
Drug: Leflunomide — tablets, 20mg, single-dose
  Other Names: ARAVA
  Arms: A
Drug: ARAVA — Tablets, 20mg, single-dose
  Other Names: Leflunomide
  Arms: B

SUMMARY:
To compare the single-dose Bioavailability of Kali and Aventis

DETAILED DESCRIPTION:
To compare the relative Bioavailability of leflunomide 20mg tablets with that of ARAVA 20mg tablets in healthy female subjects under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet all of the following criteria within 30 days prior to first drug administration(except inclusion #8)
* Healthy, surgically sterile (hysterectomy, bilateral oophorectomy) or postmenopausal (for al least 1 year)female subjects, 18 to 65 years of age(inclusive)
* Indicate non-child bearing status by one of the following criteria:

Indication of successful hysterectomy. No spontaneous menses for al least 1 year, must have luteinizing hormone (LH) and follicle stimulating hormone(FSH) levels within postmenopausal range.

Indication of successful bilateral oophorectomy.

* Body weight within 20% of the appropriate weight for the subject's height and frame (as published in the 1983 Metropolitan Life Insurance Company Scale, Statistical Bureau)
* Negative for:

HIV Hepatitis B surface antigen and Hepatitis C antibody Urine tests for drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).

Serum HCG consistent with pregnancy.

* No significant disease or clinically significant findings in a physical examination.
* No clinically significant findings in vital signs measurements and a 12-lead electrocardiogram(ECG)
* Subjects who have received leflunomide within 4 months must have an A77-1726(Metabolite) level below 0.01ug/ml and no subsequent administration of leflunomide since that test. Note: The 30 day screening limit does not apply to this inclusion criterion.
* Be informed of the nature of the study and given written consent prior to receiving any study procedures.

Exclusion Criteria:

* Subject fulfilling any of the following criteria will be excluded from the study.
* Known history or presence of any clinically significant medical condition.
* Known or suspected carcinoma.
* Known history or presence of:
* Hypersensitivity or idiosyncratic reaction to leflunomide and/or any other drug substances with similar activity.
* Alcoholism within the last 12 months.
* Drug dependence and/ or substance abuse.
* On a special diet within 4 weeks prior to drug administration(e.g. liquid, protein, raw food diet).
* Participated in another clinical trail or received an investigational product 30 days prior to drug administration.
* Donated up to 250 ml of blood in the past 45 days OR donated from 250 ml to 500 ml in the past 45 days OR donated 501 ml or more of blood in the past 56 days (based on the Canadian Blood Services guideline for blood donation).
* Requirement of any medication (prescription and/ or over-the-counter) on a routine basis, with the exception of hormonal replacement therapy, nutritional supplements and/or occasional use of common analgesics.
* Difficulty fasting or consuming the standard meals.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-12; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu Chen, Principal Investigator — Pharma Medica Research, Inc.